CLINICAL TRIAL: NCT00286312
Title: Prevention of Reperfusion Damage and Late Left Ventricular Remodelling With Atorvastatin Administered Before Reperfusion Therapy. The REPERATOR Study
Brief Title: Myocardial Infarction Size Reduction With Atorvastatin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: R&D Cardiologie (Other)
Collaborators: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RDC-2005-02
Record Dates: First submitted 2006-02-02; First posted 2006-02-03 (Estimated); Last update posted 2008-05-21 (Estimated); Status verified 2008-05

CONDITIONS: Myocardial Infarction; Reperfusion Injury
Keywords: Acute myocardial infarction; Primary angioplasty; Reperfusion damage; Atorvastatin; Placebo; Early left ventricular remodelling; Late left ventricular remodelling; Cardiac MRI; Statin; Transluminal, Percutaneous Coronary; Angioplasty
MeSH Terms: conditions — Myocardial Infarction; Reperfusion Injury | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Atorvastatin

SUMMARY:
The purpose of this study is to determine if oral atorvastatin administered just before percutaneous coronary angioplasty for acute myocardial infarction improves early and late heart function as compared to placebo.

DETAILED DESCRIPTION:
Left ventricular remodelling after a myocardial infarction refers to changes in shape and function of the infarcted and uninfarcted myocardium. Remodelling begins minutes after acute myocardial infarction and may continue for months or years, leading to dilation of the left ventricle (LV) and an increased LV volume. As studies show, LV volume strongly correlates with long-term mortality. Reperfusion after a period of ischaemia (through medication or PTCA) leads to so-called 'reperfusion injury'. This results in myocardial dysfunction and damage, which can lead to LV remodelling.

In a study where atorvastatin was administered at the onset of reperfusion infarct size was reduced. Atorvastatin led to protection of the reperfused myocardium, independently of its effects on cholesterol.

The objective is to measure the effect of atorvastatin, administered orally before reperfusion therapy by PTCA, on infarct size and microvascular reperfusion.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients (aged > 18 years) who are to undergo a primary PCI for a first acute ST elevation myocardial infarction will be asked to participate in this study.

Exclusion Criteria:

* Previous myocardial infarction
* Previous coronary artery bypass grafting (CABG)
* Cardiac rhythm is other than normal sinus rhythm.
* Electrical instability.
* The patient is in Killip class 3 or 4 of heart failure.
* Need for intra aortic balloon counterpulsation therapy
* The patient is unable to hold his/her breath for up to 20 seconds due to age or concomitant illness.
* Implanted electronic devices are present: pacemakers, internal defibrillators, ECG-registration devices, neurostimulators, implanted drug infusion devices, cochlear implants etc.
* Previous vascular surgery: aneurysm clip, carotid artery vascular clamp, aortic clips, or venous umbrella
* Prosthesis (orbital/penile, etc.)
* Spinal/intra-ventricular shunts.
* Swan-Ganz catheter; transdermal delivery systems.
* Metal fragments: eye, head, ear, skin.
* Implants held by magnets.
* Known allergy to MR contrast media
* Prior use of statins
* No PCI performed
* No recanalisation achieved

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Left ventricular end systolic volume index as measured by cine magnetic resonance imaging (MRI) at 3 month follow-up

SECONDARY OUTCOMES:
Other MRI measurements of global and regional left ventricular function
MRI measurements of infarct size at admission, 1 week, and 3 months, as well as changes in these measures between MRI investigations
Biochemical markers of infarct size
Blush grade

CONTACTS AND LOCATIONS:
Overall Officials: Benno Rensing, MD, PhD, Principal Investigator — St. Antonius Ziekenhuis Nieuwegein
Locations (2):
- Netherlands (2):
  - St. Antonius Hospital, Nieuwegein
  - University Medical Centre Utrecht, Utrecht